CLINICAL TRIAL: NCT07199530
Title: Association Between Elevated Plasma D Dimer in Adult Community- Acquired Pneumonia Patients and Severity of Inflammatory Response and Survival
Brief Title: Association Between Plasma D Dimer in Adult CAP and Severity of Inflammatory Response and Survival
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, hieba gamal ezz-elragal awad, assistant professor, Ain Shams University
Other Study IDs: FAMSU R 135/2025
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: D-dimer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- only one group which will include patients with CAP to take a blood samplr for d dimer
  Interventions: Other: Blood Product

INTERVENTIONS:
Other: Blood Product — blood sample for d dimer

SUMMARY:
This is an observational study aiming to investigate the association between elevated plasma D-dimer levels and the inflammatory response, as well as the impact on survival in adult patients with community acquired pneumonia.

the study participants will be subjected to sampling for D dimer and calculation of CURB 65 score. this aims to find the relation between them

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is a common and potentially life-threatening infection that affects millions of individuals worldwide each year.

D-dimer is a fibrin degradation product that is elevated in many conditions associated with inflammation and coagulation activation, including pneumonia.

This is an observational study including a minimum of 50 patients with CAP

Patients who will be admitted at Chest department, or coming to the outpatient clinic Ain-Shams University Hospitals with CAP and have the following inclusions:

1. age ≥18 years
2. diagnosis of CAP based on clinical symptoms, laboratory findings, and radiological evidence.
3. Did not have any clinical or radiological signs suggesting Covid pneumonia Exclusion criteria Patients with a history of coagulation disorders, cancer, or other chronic diseases, or refusal to participate.

All patients will be subjected to the following: -

1. Full medical history, demographics
2. Thorough clinical examination.
3. laboratory values (including white blood cell count, CRP, and D-dimer), With pre and post sample known precautions (8).
4. Radiological findings (CXR).
5. Severity of illness (based on the CURB-65 score).

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be admitted at Chest department, or coming to the outpatient clinic Ain-Shams University Hospitals with CAP and have the following inculsions:

  1. age ≥18 years
  2. diagnosis of CAP based on clinical symptoms, laboratory findings, and radiological evidence.

Exclusion Criteria:

* Patients with a history of coagulation disorders, cancer, or other chronic diseases, or refusal to participate.
* patients who have any clinical or radiological signs suggesting Covid pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the participant is those patients with CAP WHO will meet the inclusion criteria previously mentioned
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
find the association between plasma D dimer level and severity of CAP | in 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
to save patients DATA